CLINICAL TRIAL: NCT05784597
Title: A Phase I Study to Evaluate the Safety and Dosimetry of 68Ga-labelled OncoFAP Derivatives in Patients with Solid Tumors
Brief Title: A Study to Evaluate the Safety and Dosimetry of 68Ga-labelled OncoFAP Derivatives in Solid Tumors
Acronym: FAPrimo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PH-FAPGA-01/22
Record Dates: First submitted 2022-12-15; First posted 2023-03-27 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Colorectal Cancer; Oesophageal Cancer; Pancreas Adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are divided into two cohorts:
  * Cohort A: 3 female + 3 male patients with a primary tumor only
  * Cohort B: patients with a primary tumor and/or advanced/metastatic disease with a quantifiable number of lesions (6 - 14 patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): 3 female + 3 male patients with a primary tumor only
  Interventions: Drug: [68Ga]Ga-OncoFAP administration
- Cohort B (Experimental): Patients with a primary tumor and/or advanced/metastatic disease with a quantifiable number of lesions
  Interventions: Drug: [68Ga]Ga-OncoFAP administration

INTERVENTIONS:
Drug: [68Ga]Ga-OncoFAP administration — All patients will receive a single intravenous bolus administration of 250 MBq (225 - 275 MBq)

SUMMARY:
The primary objectives of this trial are to evaluate the safety and dosimetry of [68Ga]Ga-OncoFAP for detection/imaging of solid tumors.

DETAILED DESCRIPTION:
Phase I, multicenter study in patients with a confirmed diagnosis of solid tumor among breast cancer, colorectal cancer, oesophageal cancer and pancreatic adenocarcinoma, requiring clinical staging for nodal staging and/or metastatic disease (based on institutional practice and risk stratification). All patients will receive a single intravenous bolus administration of 250 MBq (225 - 275 MBq). [68Ga]Ga-OncoFAP biodistribution, PK, and dosimetry of [68Ga]Ga-OncoFAP will be assessed based on a series of PET/CT scans, blood and urine sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of breast cancer, colorectal cancer, oesophageal cancer and pancreatic adenocarcinoma. Confirmation by histopathology is required for breast, colorectal and oesophageal cancer. For pancreatic adenocarcinoma, confirmation by histopathology or cytology obtained by endoscopic ultrasound is accepted.
2. Requirement for diagnostic imaging or imaging performed within 4 weeks prior to the [68Ga]Ga-OncoFAP-PET/CT scan for staging.
3. Male or non-pregnant and non-breastfeeding female.
4. For female patients: negative serum pregnancy test for women of childbearing potential* (WOCBP).

   WOCBP must agree to use, from the screening to six months following the study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.
5. For male patients: male subject able to father children must agree to practice effective contraception for three months starting from the study drug administration.
6. Age 18 - 75
7. ECOG ≤ 1
8. Patient must not have any concomitant infections or active concomitant disease.
9. Life expectancy of more than 12 weeks.
10. Ability to undergo imaging study procedures.
11. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
12. Willingness and ability to comply with the scheduled visits, plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).

Exclusion Criteria:

1. Chronically impaired renal function as expressed by creatinine clearance < 60 mL/min or serum creatinine > 1.5 x ULN.
2. Presence of active hepatitis.
3. Presence of significant cardiac disorders (congestive heart failure, NYHA class III-IV, myocardial infarction within one year prior to study entry, uncontrolled hypertension, or arrhythmia).
4. Pregnant or breastfeeding during participation in the study.
5. Any concomitant condition which in the opinion of investigators makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
6. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of the study drug. Minimally invasive procedures such as biopsies are not considered as exclusion criteria.
7. Serious, non-healing wound, ulcer, or bone fracture.
8. Allergy to study medication or excipients in study medication.
9. Any anti-cancer therapy (e.g. cytotoxic chemotherapy, immunotherapy, radiation, surgery, etc.) within 3 weeks before [68Ga]Ga-OncoFAP-PET/CT scan
10. Subject has received, or is scheduled to receive, another investigational medicinal product (IMP) from 1 month before [68Ga]Ga-OncoFAP injection to end of study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Safety (AE) | Throughout study, until a maximum of 8 days after the completion of each patient
  Safety of administration of 68Ga-OncoFAP, assessed based on Common Toxicity Criteria (CTCAE version 5.0)
Cohort A: Dosimetry - Effective dose equivalent (mSv) | Assessed on day 1
  Effective dose equivalent (mSv) of normal organs following administration of a single dose of [68Ga]Ga-OncoFAP, for patients in cohort A
Cohort A: Dosimetry - Absorbed doses (mGy) | Assessed on day 1
  Absorbed doses (mGy) of normal organs following administration of a single dose of [68Ga]Ga-OncoFAP, for patients in cohort A

SECONDARY OUTCOMES:
Biodistribution profile: SUVmax | Assessed on day 1
  Uptake of [68Ga]Ga-OncoFAP in terms of SUVmax
Biodistribution profile: SUVmean | Assessed on day 1
  Uptake of [68Ga]Ga-OncoFAP in terms of SUVmean
Biodistribution profile: SUVsd | Assessed on day 1
  Uptake of [68Ga]Ga-OncoFAP in terms of SUVsd
PK | Assessed on day 1
  Pharmacokinetics of [68Ga]Ga-OncoFAP based on measurement of residual radioactivity in the blood over time [MBq/mL
Excretion | Assessed on day 1
  Metabolism and excretion of [68Ga]Ga-OncoFAP based on radioactivity measurements on urine collected at defined timepoints
Immunopathology staining | Assessed on day 1
  Correlation of [68Ga]Ga-OncoFAP uptake with immunopathology staining if and when surgical or biopsy specimen are available
Lesion detection rate | Assessed on day 1
  Lesion detection rate compared to standard imaging

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Istituto Nazionale dei Tumori | Fondazione IRCCS, Milan, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - IRCCS San Raffaele, Milan